CLINICAL TRIAL: NCT03017352
Title: Meal-time Administration of Exenatide for Glycaemic Control in Type 1 Diabetic Cases: A Randomised, Placebo-controlled Trial
Brief Title: Meal-time Administration of Exenatide for Glycaemic Control in Type 1 Diabetic Cases
Acronym: MAG1C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Filip Krag Knop (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Filip Krag Knop, Professor, MD, PhD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Eudract-nr.: 2016-001365-92
Record Dates: First submitted 2017-01-02; First posted 2017-01-11 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Exenatide; Incretins; GLP-1; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Exenatide 10 mikrogram, thrice daily, subcutaneous injection prior to main meals, 6 months.
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): Placebo, thrice daily, subcutaneous injection prior to main meals, 6 months.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Exenatide
  Other Names: Byetta
  Arms: Intervention
Drug: Placebos
  Arms: Placebo

SUMMARY:
Patients with type 1 diabetes (T1D) depend on insulin therapy as substitution for the lack of endocrine insulin production due to an autoimmune destruction of beta-cells in the pancreatic inslets. Insulin therapy is based on long lasting basal insulin for controlling fasting plasma glucose, and short lasting mealtime insulin for the postprandial plasma glucose. The long term efficacy of this treatment is measured in glycated haemoglobin A1c (HbA1c) of <7.0% as the treatment goal.

Intensive insulin therapy is associated with side effects such as hypoglycaemia, weight gain, and unwanted exaggerated excursions in PPG. This may ultimately affect treatment compliance.

The abovementioned problems associated with insulin treatment in T1D can also be seen in insulin-treated patients with type 2 diabetes (T2D). However, in T2D the combination of insulin with glucagon-like peptide-1 (GLP-1) receptor agonist (RA) has proven effective in reducing the weight gain and insulin dose in insulin-treated patients with T2D without exacerbating the risk of hypoglycaemia.

Exenatid is a short lasting GLP-1RA approved for treatment in T2D, and the investigators intend to evaluate it in a randomized, controlled trial as add-on therapy to standard insulin therapy for patients with T1D.

The investigators hypothesise that the add-on of exenatide to insulin therapy in patients with T1D will reduce insulin requirements, glycaemic excursions and body weight and improve glycaemic control without increasing the risk of hypoglycaemia.

ELIGIBILITY:
Inclusion Criteria:

* T1D according to WHO criteria with duration of ≥1 year
* Age ≥18 years
* BMI >22.0 kg/m2
* HbA1c >7.5% and <10.0% at visit 0 (screening)
* Able to count carbohydrates

Exclusion Criteria:

* Insulin pump treatment
* Hypoglycaemia unawareness (inability to register low blood glucose)
* Diabetic gastroparesis
* Compromised kidney function (eGFR <60 ml/min/1.73m2, dialysis or kidney transplantation)
* Liver disease with elevated plasma alanine aminotransferase (ALT) > three times the upper limit of normal (measured at visit 0 with the possibility of one repeat analysis within a week, and the last measured value as being conclusive)
* History of acute and/or chronic pancreatitis
* Subjects with personal or family history of medullary carcinoma or MEN syndrome
* Inflammatory bowel disease
* Cancer unless in complete remission for >5 years
* Proliferative retinopathy
* Other concomitant disease or treatment that according to the investigator's assessment makes the patient unsuitable for study participation
* Alcohol/drug abuse
* Fertile women not using chemical (tablet/pill, depot injection of progesterone, subdermal gestagen implantation, hormonal vaginal ring or transdermal hormonal patch) or mechanical (spirals) contraceptives
* Pregnant or nursing women
* Known or suspected hypersensitivity to trial product or related products
* Receipt of an investigational drug within 30 days prior to visit 0
* Simultaneous participation in any other clinical intervention trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-12; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months
  Change in HbA1c from baseline to end of study (time 6 months)

SECONDARY OUTCOMES:
adverse events (including hypoglycaemic episodes) | 6 months
changes in insulin dosage | 6 months
changes in body weight | 6 months
changes in BMI | 6 months
changes in body composition | 6 months
  DXA scan measuring bonemineral density
changes in body composition | 6 months
  DXA scan measuring lean mass
changes in body composition | 6 months
  DXA scan measuring fat mass
changes in fasting plasma glucose | 6 months
changes in post prandial plasma glucose | 6 months
changes in fasting plasma levels of C-peptide | 6 months
Quality of life self reported | 6 months
  Quality of Life Questionaire
Treatment satisfaction | 6 months
  Diabetes treatment satisfactory questionnaire status version
Treatment satisfaction | 6 months
  Diabetes treatment satisfactory questionnaire change version
dietary patterns | 6 months
  Food frequency questionaire three times during the intervention
HDL (High Density Lipoprotein) | 6 months
LDL (Low Density Lipoprotein) | 6 months
VLDL (Very Low Density Lipoprotein) | 6 months
total cholesterol | 6 months
triglycerides | 6 months
proBNP (Pro-Brain Natriuretic Peptide) | 6 months
hsCRP (High-Sensitivity C-Reactive Protein) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Capital Region, Denmark

REFERENCES:
- [Background] Johansen NJ, Dejgaard TF, Lund A, Vilsboll T, Andersen HU, Knop FK. Protocol for Meal-time Administration of Exenatide for Glycaemic Control in Type 1 Diabetes Cases (The MAG1C trial): a randomised, double-blinded, placebo-controlled trial. BMJ Open. 2018 Jun 27;8(6):e021861. doi: 10.1136/bmjopen-2018-021861. PMID 29950475
- [Derived] Johansen NJ, Dejgaard TF, Lund A, Schluntz C, Frandsen CS, Forman JL, Wewer Albrechtsen NJ, Holst JJ, Pedersen-Bjergaard U, Madsbad S, Vilsboll T, Andersen HU, Knop FK. Efficacy and safety of meal-time administration of short-acting exenatide for glycaemic control in type 1 diabetes (MAG1C): a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2020 Apr;8(4):313-324. doi: 10.1016/S2213-8587(20)30030-9. Epub 2020 Mar 2. PMID 32135138